CLINICAL TRIAL: NCT02882724
Title: Effect Aquatic Exercise Training on Patients With Multiple Sclerosis
Brief Title: Changes in Speed, Endurance and Balance in Women Patients With Multiple Sclerosis After 4 & 8 Weeks of Aquatic Exercise Training
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Isfahan (Other)
Responsible Party: Principal Investigator, Prof.Mehdi Kargarfard, Principal Investigator, University of Isfahan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201527921IR
Record Dates: First submitted 2016-08-15; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis; Aquatic; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

ARMS (2):
- Exercise training (Experimental)
  Interventions: Behavioral: Exercise
- Control (Experimental): Control group did not do any exercise training.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise — 8-week aquatic exercise training program
  Arms: Exercise training
Behavioral: Control — Control group did not do the exercise training.
  Arms: Control

SUMMARY:
Background: It has been shown that adults with Multiple sclerosis (MS) have less leg strength than their peers, as well as impaired balance, which has led to an increased prevalence of falls in this population.The purpose of this study was to assess the effects of 8-weeks aquatic exercise training in balance, endurance and speed in women with MS.

Methods: In this semi-experimental study, 32 women with clinically-definite relapsing-remittent MS who were registered through the Isfahan MS association volunteered for this study. They randomly selected an aquatic exercise (n = 17) and control (n = 15) groups. Aquatic exercise group completed a 8-week aquatic exercise training program consisted of three sessions per week, each session lasting 45 to 60 minutes 50 to 75 percent of their maximum heart rate reserve on 20-25 degree centigrade's, whereas the control group was instructed to maintain their current lifestyle. The balance of angry was surveyed with using of Berg analyze, speed and endurance 6 minutes walking test before starting of exercise program and after 4 weeks and at the end of 8 weeks was analyzed. The obtained data's were analyzed using analysis of variance with repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* All women diagnosis of clinically or laboratory supported MS, a minimum time of two years since the diagnosis was made, no relapse within the 4 weeks preceding baseline, ability to participate in regular exercise sessions.

Exclusion Criteria:

* Patients were excluded from the study if they had a relapse during the intervention period, and had a disease preventing their participation (e.g. cardiovascular, respiratory or skeletal diseases).

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Effect of exercise on balance was surveyed with using of Berg analyze | up to 8 weeks

SECONDARY OUTCOMES:
Effect of exercise on speed was measured by walking test | Up to 8 weeks
Effect of exercise on endurance was measured by walking test | Up to 8 weeks

REFERENCES:
- [Derived] Kargarfard M, Shariat A, Ingle L, Cleland JA, Kargarfard M. Randomized Controlled Trial to Examine the Impact of Aquatic Exercise Training on Functional Capacity, Balance, and Perceptions of Fatigue in Female Patients With Multiple Sclerosis. Arch Phys Med Rehabil. 2018 Feb;99(2):234-241. doi: 10.1016/j.apmr.2017.06.015. Epub 2017 Jul 20. PMID 28735720